CLINICAL TRIAL: NCT06975735
Title: Does the Transversalis Fascia Plane Block Work Better Than the Transversus Abdominis Plane Block for Relieving Pain After a Robotic-assisted Partial Prostatectomy?
Brief Title: Does the TAP Block Work Better Than the TFP Block for Relieving Pain
Acronym: Tapblock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kudret Dogru, Prof. Dr. (MD), TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/184
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pain
Keywords: prostatectomy, pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAP Group (Active Comparator): Receiving TAP 20 ml bupivacaine 0.25%
  Interventions: Procedure: TAP Plane Block
- TFP Group (Active Comparator): Receiving TFP 20 ml bupivacaine 0.25%
  Interventions: Procedure: TFP Block
- Control Group (No Intervention): Not receiving TAP or TFP

INTERVENTIONS:
Procedure: TAP Plane Block — The transversus abdominis plane block (TAPB) is a technically simple and safe form of regional anesthesia that can provide effective analgesia for 12 hours in patients with acute postoperative pain
  Other Names: TAP Block
  Arms: TAP Group
Procedure: TFP Block — The transversalis fascia plane block (TAPB) is a technically simple and safe form of regional anesthesia that can provide effective analgesia for 12 hours in patients with acute postoperative pain
  Arms: TFP Group

SUMMARY:
Regional anesthetics, nerve blocks, and interfascial blocks are becoming more common in many types of surgery to help with pain after surgery. Most clinicians concur with the importance of reducing postoperative pain scores and facilitating early discharge. The transversalis fascia plane block (TFP) and transversus abdominis plane block (TA), which are done from the side of the abdomen, have been proven to be very useful in surgeries related to women's health, weight loss, and the colon. Research on the effectiveness of both procedures in robot-assisted laparoscopic prostatectomies (RALP) is insufficient. The aim was to see if using a transversalis fascia plane block (TFP) or a transversus abdominal plane (TAP) block with 0.25% bupivacaine helped reduce pain, speed up recovery, and shorten hospital stays for men undergoing robot-assisted radical prostatectomy (RALP).

DETAILED DESCRIPTION:
Regional anesthetics, nerve blocks, and interfascial blocks are becoming more common in many types of surgery to help with pain after surgery. Most clinicians concur with the importance of reducing postoperative pain scores and facilitating early discharge. The transversalis fascia plane block (TFP) and transversus abdominis plane block (TA), which are given from the side of the abdomen, have been found to be very useful in surgeries related to women's health, weight loss, and the colon. Research shows that both procedures are ineffective in robot-assisted laparoscopic prostatectomies (RALP).

In this study, doctors will start general anesthesia using propofol and rocuronium as usual and keep it going with a mix of 4-6% desflurane with oxygen, remifentanil, and rocuronium given through an IV.

All procedures will be conducted within the framework of an observational clinical research protocol, and patients will not be subjected to any procedures outside of routine practices.

Before starting the study, patients will be thoroughly informed, and their written consent will be obtained. The study is planned to start in May 2025.

Patients will be examined in the anesthesia outpatient clinic for preoperative evaluation. Demographic data (age, gender, ASA score, height, weight, BMI, and comorbidities) will be recorded in the preoperative patient evaluation form.

Standard monitoring included invasive and non-invasive blood pressure measurements, electrocardiography (ECG), and pulse oximetry. During anesthesia, balanced IV fluid replacement will be provided through a 20-G arterial and three 18-G intravenous cannulas. The patient will be placed in a supine and Trendelenburg surgical position.

This study has been planned as prospective and observational in nature. In this study, patients who undergo robotic-assisted partial prostatectomy at our hospital and will receive a transversalis fascia plane block (TFPB) or transversus abdominis plane (TAP) block as a standard practice for postoperative pain relief will be followed. Patients who choose not to have these blocks during the pre-surgery information will be placed in the control group and will receive pain relief in the same manner. The control group will include patients who refuse these block applications during preoperative information, and they will receive postoperative analgesia in the same manner.

Which block technique will be applied will be determined entirely by the clinician's decision regarding these cases and the patient's characteristics, and no randomization, intervention, or guidance will be carried out by the researchers.

Groups: 1-Group TFP, 2-Group TAP, 3-Group Control Postoperative analgesic efficacy will be evaluated at 1, 6, and 24 hours. Postoperative pain will be evaluated both at rest and during coughing using a 0-10 point visual analog scale (VAS). As usual, morphine (5 mg i.v.) and paracetamol (1000 mg i.v.) will be provided and recorded as rescue analgesia for pain scores exceeding 3/10 during rest or coughing.

The time of the patients' first standing and walking will be recorded, and the surgeon's satisfaction with postoperative patient comfort will be scored as 1-Excellent, 2-Good, or 3-Poor.

Among the groups, VAS scores, rescue analgesics, postoperative ambulation time, postoperative satisfaction scores (patient and surgeon perspective), and complications such as possible nausea, vomiting, and hypotension will be compared.

The researchers used G Power software to analyze the study's strength before it started, focusing on the average Visual Analog Score in each group, which is the key factor for their main hypothesis. Based on earlier research, they determined that an effect size of 0.35 is important for clinical significance, and using the ANOVA test, they found that they need at least 36 patients in each group, which adds up to 108 patients in total. With this calculation, the power of the study is based on 0.90 and a significance level (α) of 0.05.

The data will be evaluated for normal distribution using the Shapiro-Wilk test and for homogeneity using the Levene test. For normally distributed, homogeneous data, ANOVA and post hoc Tukey tests will be used, while Kruskal-Wallis and chi-square tests will be used for categorical and non-normally distributed data. When necessary, the Bonferroni correction will be applied. For multiple comparisons, those with a p-value < 0.05 will be considered statistically significant. All statistical analyses will be conducted using JAMOVI version 2.6.19 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I or II
* Having regular preoperative visits

Exclusion Criteria:

1. Patients classified as ASA III or IV,
2. Patients with coagulopathy
3. Those with a history of allergies
4. Significant Cardiac Disorders (Coronary Artery Disease, Arrhythmia, Electrocardiography Anomaly, Heart Failure, etc.)

1. Those with bleeding diathesis and those receiving anticoagulant therapy 2. Those with a history of carotid artery stenosis, 3. Cardiovascular disease, 4. Hipertansiyon, 5. Chronic obstructive pulmonary disease, 6. Patients with a heart rhythm outside the sinus 7. Patients with a history of cerebrovascular disease 8. Alcoholism or psychiatric illness 9. Those with diabetes, 10. Contraindicated for TAP and TFP Block 11. Those with drug allergies

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only male patients
Enrollment: 108 (Actual)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Reducing patient-controlled analgesic consumption | From the patient's anesthesia induction in the operating room to the postoperative 24. hours
  The time to first analgesic request in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Kudret Doğru, Prof. Dr., Study Director — TC Erciyes University
Locations (1):
- Kudret Doğru, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dal Moro F, Aiello L, Pavarin P, Zattoni F. Ultrasound-guided transversus abdominis plane block (US-TAPb) for robot-assisted radical prostatectomy: a novel '4-point' technique-results of a prospective, randomized study. J Robot Surg. 2019 Feb;13(1):147-151. doi: 10.1007/s11701-018-0858-6. Epub 2018 Jul 28. PMID 30056612
- [Background] Cacciamani GE, Menestrina N, Pirozzi M, Tafuri A, Corsi P, De Marchi D, Inverardi D, Processali T, Trabacchin N, De Michele M, Sebben M, Cerruto MA, De Marco V, Migliorini F, Porcaro AB, Artibani W. Impact of Combination of Local Anesthetic Wounds Infiltration and Ultrasound Transversus Abdominal Plane Block in Patients Undergoing Robot-Assisted Radical Prostatectomy: Perioperative Results of a Double-Blind Randomized Controlled Trial. J Endourol. 2019 Apr;33(4):295-301. doi: 10.1089/end.2018.0761. Epub 2019 Jan 31. PMID 30484332